CLINICAL TRIAL: NCT03987074
Title: A Proof of Concept, Open-Label Study Evaluating the Safety, Tolerability, and Efficacy of Monotherapy and Combination Regimens in Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Safety, Tolerability, and Efficacy of Monotherapy and Combination Regimens in Participants With Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-454-5533
Record Dates: First submitted 2019-06-12; First posted 2019-06-14 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — semaglutide; firsocostat; cilofexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Semaglutide (Experimental): Semaglutide 0.24 mg - 2.4 mg (dose escalated over 16 weeks) for 24 weeks
  Interventions: Drug: Semaglutide
- Semaglutide + Firsocostat 20 mg (Experimental): Semaglutide 0.24 mg - 2.4 mg (dose escalated over 16 weeks) + firsocostat 20 mg for 24 weeks
  Interventions: Drug: Semaglutide; Drug: Firsocostat
- Semaglutide + Cilofexor 30 mg (Experimental): Semaglutide 0.24 mg - 2.4 mg (dose escalated over 16 weeks) + cilofexor 30 mg for 24 weeks
  Interventions: Drug: Semaglutide; Drug: Cilofexor
- Semaglutide + Cilofexor 100 mg (Experimental): Semaglutide 0.24 mg - 2.4 mg (dose escalated over 16 weeks) + cilofexor 100 mg for 24 weeks
  Interventions: Drug: Semaglutide; Drug: Cilofexor
- Semaglutide + Firsocostat 20 mg + Cilofexor 30 mg (Experimental): Semaglutide 0.24 mg - 2.4 mg (dose escalated over 16 weeks) + firsocostat 20 mg + cilofexor 30 mg for 24 weeks
  Interventions: Drug: Semaglutide; Drug: Firsocostat; Drug: Cilofexor

INTERVENTIONS:
Drug: Semaglutide — Solution administered subcutaneously with pre-filled PDS290 pen-injector once weekly
Drug: Firsocostat — Tablets administered orally once daily
  Other Names: GS-0976
  Arms: Semaglutide + Firsocostat 20 mg; Semaglutide + Firsocostat 20 mg + Cilofexor 30 mg
Drug: Cilofexor — Tablets administered orally once daily
  Other Names: GS-9674
  Arms: Semaglutide + Cilofexor 100 mg; Semaglutide + Cilofexor 30 mg; Semaglutide + Firsocostat 20 mg + Cilofexor 30 mg

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of study drug(s) in participants with nonalcoholic steatohepatitis (NASH).

ELIGIBILITY:
Key Inclusion Criteria:

* Historical liver biopsy consistent with NASH with stage 2-3 fibrosis according to NASH Clinical Research Network (CRN) classification OR clinical diagnosis of nonalcoholic fatty liver disease and screening FibroTest, magnetic resonance imaging - proton density fat fraction (MRI-PDFF), and FibroScan
* Screening laboratory parameters, as determined by central laboratory:

  * Alanine aminotransferase (ALT) ≤ 5 x upper limit of the normal range (ULN)
  * Estimated glomerular filtration rate (eGFR) ≥ 30 milliliter/minute (mL/min), as calculated by the Modification of Diet in Renal Disease (MDRD) study equation
  * HbA1c ≤ 9.5%
  * International normalized ratio (INR) ≤ 1.2, unless due to therapeutic anti-coagulation therapy
  * Platelet count ≥ 100,000/μL
  * Total bilirubin < 1.3 x ULN unless alternate etiology such as Gilbert's syndrome present
  * Calcitonin ≤ 100 ng/L
* Body Mass Index (BMI) > 23 kg/m^2 and body weight of > 60 kg

Key Exclusion Criteria:

* Any historical liver biopsy consistent with cirrhosis
* Any history of decompensated liver disease, including ascites, hepatic encephalopathy, or variceal bleeding
* Other causes of liver disease, including but not limited to: alcoholic liver disease, hepatitis B, hepatitis C, autoimmune disorders (eg, primary biliary cholangitis (PBC), primary sclerosing cholangitis (PSC), autoimmune hepatitis), drug-induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1-antitrypsin deficiency requiring treatment
* History of liver transplantation
* History of hepatocellular carcinoma
* History of pancreatitis (acute or chronic)
* Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma
* Treatment with glucagon-like peptide-1 receptor agonists (GLP-1 RA) in the period from 90 days prior to the date of the Screening Visit
* Individuals on antidiabetic medications must be on a stable dose for at least 90 days prior to the date of the Screening Visit and in the period between the date of the Screening Visit and Enrollment (Day -14)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (18):
- United States (18):
  - Institute for Liver Health - Arizona Liver Health, Chandler, Arizona
  - Southern California Research Centers, Coronado, California
  - University of California San Diego (UCSD), La Jolla, California
  - Ruane Clinical Research Group, Inc, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Medical Associates Research Group, San Diego, California
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - Northwell Health, Manhasset, New York
  - Gastro One, Huntersville, North Carolina
  - University Gastroenterology, Providence, Rhode Island
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - American Research Corporation, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alkhouri N et al. Safety and Efficacy of Combination Therapies Including Semaglutide, Cilofexor, and Firsocostat in Patients with NASH [accepted for oral presentation]. American Association for the Study of Liver Diseases (AASLD); 2020; Virtual.
- [Derived] Alkhouri N, Herring R, Kabler H, Kayali Z, Hassanein T, Kohli A, Huss RS, Zhu Y, Billin AN, Damgaard LH, Buchholtz K, Kjaer MS, Balendran C, Myers RP, Loomba R, Noureddin M. Safety and efficacy of combination therapy with semaglutide, cilofexor and firsocostat in patients with non-alcoholic steatohepatitis: A randomised, open-label phase II trial. J Hepatol. 2022 Sep;77(3):607-618. doi: 10.1016/j.jhep.2022.04.003. Epub 2022 Apr 16. PMID 35439567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 29 July 2019. The last study visit occurred on 13 July 2020.
Pre-assignment Details: 209 participants were screened. 109 participants were enrolled. 1 participant was enrolled but was not randomized and was not included in the analysis.
Groups:
- Semaglutide: Participants received semaglutide 0.24 mg - 2.4 mg (dose escalated over 16 weeks) subcutaneously with prefilled PDS290 pen-injector once weekly for 24 weeks.
- Semaglutide + Firsocostat 20 mg: Participants received semaglutide 0.24 mg - 2.4 mg (dose escalated over 16 weeks) subcutaneously with prefilled PDS290 pen-injector once weekly for 24 weeks + firsocostat 20 mg tablet orally once daily with or without food for 24 weeks.
- Semaglutide + Cilofexor 30 mg: Participants received semaglutide 0.24 mg - 2.4 mg (dose escalated over 16 weeks) subcutaneously with prefilled PDS290 pen-injector once weekly for 24 weeks + cilofexor 30 mg tablet orally once daily with or without food for 24 weeks.
- Semaglutide + Cilofexor 100 mg: Participants received semaglutide 0.24 mg - 2.4 mg (dose escalated over 16 weeks) subcutaneously with prefilled PDS290 pen-injector once weekly for 24 weeks + cilofexor 100 mg tablet orally once daily with or without food for 24 weeks.
- Semaglutide + Firsocostat 20 mg + Cilofexor 30 mg: Participants received semaglutide 0.24 mg - 2.4 mg (dose escalated over 16 weeks) subcutaneously with prefilled PDS290 pen-injector once weekly for 24 weeks + firsocostat 20 mg tablet orally once daily + cilofexor 30 mg tablet orally once daily with or without food for 24 weeks.
Period: Overall Study
Arm/Group | Semaglutide | Semaglutide + Firsocostat 20 mg | Semaglutide + Cilofexor 30 mg | Semaglutide + Cilofexor 100 mg | Semaglutide + Firsocostat 20 mg + Cilofexor 30 mg
Started | 21 | 22 | 22 | 22 | 21
Completed | 18 | 20 | 21 | 18 | 19
Not Completed | 3 | 2 | 1 | 4 | 2
Not completed — Withdrew Consent | 1 | 1 | 0 | 2 | 1
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0
Not completed — Investigator's Discretion | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Semaglutide + Firsocostat 20 mg | Semaglutide + Cilofexor 30 mg | Semaglutide + Cilofexor 100 mg | Semaglutide + Firsocostat 20 mg + Cilofexor 30 mg | Total
Number analyzed (Participants) | 21 | 22 | 22 | 22 | 21 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10.4) | 52 (12.6) | 51 (10.9) | 54 (10.8) | 53 (11.4) | 53 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 16 | 13 | 15 | 74
  Male | 6 | 7 | 6 | 9 | 6 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 1 | 4
  Asian | 2 | 2 | 2 | 1 | 0 | 7
  Black | 1 | 0 | 1 | 1 | 0 | 3
  White | 17 | 19 | 18 | 19 | 19 | 92
  Other | 0 | 1 | 0 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 13 | 10 | 17 | 15 | 10 | 65
  Hispanic or Latino | 8 | 12 | 5 | 7 | 11 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events (TEAEs) were defined as, any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug or any AEs leading to premature discontinuation of study drug. Participants were assessed for AEs according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: First dose date up to Week 24 plus 30 days
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Semaglutide | Semaglutide + Firsocostat 20 mg | Semaglutide + Cilofexor 30 mg | Semaglutide + Cilofexor 100 mg | Semaglutide + Firsocostat 20 mg + Cilofexor 30 mg
Number analyzed (Participants) | 21 | 22 | 22 | 22 | 21
percentage of participants | 81.0 | 86.4 | 81.8 | 72.7 | 90.5

2. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities, defined as values that increase at least one toxicity grade from baseline at any time post-baseline up to and including the date of last dose of study drug plus 30 days, were summarized by treatment group. Graded laboratory abnormalities were defined using the grading scheme in the CTCAE 5.0.
Time Frame: First dose date up to 24 weeks plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Semaglutide | Semaglutide + Firsocostat 20 mg | Semaglutide + Cilofexor 30 mg | Semaglutide + Cilofexor 100 mg | Semaglutide + Firsocostat 20 mg + Cilofexor 30 mg
Number analyzed (Participants) | 21 | 22 | 22 | 22 | 21
percentage of participants
  Grade 1 | 61.9 | 63.6 | 36.4 | 50.0 | 66.7
  Grade 2 | 23.8 | 22.7 | 31.8 | 18.2 | 9.5
  Grade 3 | 0.0 | 4.5 | 0.0 | 0.0 | 0.0
  Grade 4 | 0.0 | 0.0 | 0.0 | 9.1 | 0.0

ADVERSE EVENTS:
Time Frame: First dose date up to 24 weeks plus 30 days
Description: The Safety Analysis Set included participants who received at least 1 dose of study drug
Groups:
- Semaglutide + Cilofexor 100 mg: Semaglutide + Cilofexor 100 mg Participants received semaglutide 0.24 mg - 2.4 mg (dose escalated over 16 weeks) subcutaneously with prefilled PDS290 pen-injector once weekly for 24 weeks + cilofexor 100 mg tablet orally once daily with or without food for 24 weeks.
Arm/Group | Semaglutide | Semaglutide + Firsocostat 20 mg | Semaglutide + Cilofexor 30 mg | Semaglutide + Cilofexor 100 mg | Semaglutide + Firsocostat 20 mg + Cilofexor 30 mg
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/22 | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/22 | 0/22 | 1/22 | 0/21
Other Adverse Events (participants affected / at risk) | 16/21 | 17/22 | 18/22 | 13/22 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Semaglutide (N=21) | Semaglutide + Firsocostat 20 mg (N=22) | Semaglutide + Cilofexor 30 mg (N=22) | Semaglutide + Cilofexor 100 mg (N=22) | Semaglutide + Firsocostat 20 mg + Cilofexor 30 mg (N=21)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Semaglutide (N=21) | Semaglutide + Firsocostat 20 mg (N=22) | Semaglutide + Cilofexor 30 mg (N=22) | Semaglutide + Cilofexor 100 mg (N=22) | Semaglutide + Firsocostat 20 mg + Cilofexor 30 mg (N=21)
Vision blurred (Eye disorders) | 0 | 0 | 2 | 0 | 0
Visual impairment (Eye disorders) | 0 | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 5 | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 5 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 3 | 8 | 6 | 14
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 6
Early satiety (General disorders) | 1 | 3 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 3 | 1 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 2 | 1
Weight decreased (Investigations) | 0 | 0 | 2 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4 | 6 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 3 | 2 | 0
Headache (Nervous system disorders) | 1 | 3 | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT03987074/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT03987074/SAP_001.pdf